CLINICAL TRIAL: NCT02863848
Title: Effect of Inulin-type Fructans on Constipated Children. Pilot Study.
Brief Title: Effect of Inulin-type Fructans on Constipated Children.
Acronym: CONSTICHILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Beneo GmbH (Industry)
Responsible Party: Principal Investigator, Dr. Joaquin Escribano, Head of the Paediatrics, Nutrition and Human Development Research Unit Universitat Rovira i Virgili - IISPV, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONSTICHILD
Record Dates: First submitted 2016-04-04; First posted 2016-08-11 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin 2g, twice per day, 6 weeks
  Interventions: Dietary Supplement: Placebo
- Inulin-type fructans (Active Comparator): Orafti inulin-type fructans 2g, twice per day, 6 weeks
  Interventions: Dietary Supplement: OraftiR inulin-type fructans

INTERVENTIONS:
Dietary Supplement: OraftiR inulin-type fructans
  Arms: Inulin-type fructans
Dietary Supplement: Placebo — maltodextrin
  Arms: Placebo

SUMMARY:
The main objective of this Pilot study was to assess the beneficial effects of a daily supplementation with Orafti inulin-type fructans in 2-5 year old constipated children The study is primary aimed to develop a feasibility study to assess the beneficial effect of inulin-type fructans in the described population with regard to the adequate criteria for a larger trial. Secondary objectives are to obtain data about the feasibility of the protocol (as pilot study). To obtain data useful to perform sample size calculations for a big study designed specifically to investigate the beneficial effect of inulin-type fructans in the treatment of constipated children.

Study design and subjects: Double-blind, randomized, placebo-controlled parallel group trial; where 2-5 year-old constipated children received inulin-type fructans or the same amount of placebo (maltodextrin) during 6 weeks. The study protocol was approved by the local Ethical Committees.

Outcomes: primary outcome was stool consistency. Secondary outcomes were: stool frequency, gastrointestinal symptoms (abdominal pain and pain during defecation), additional medication required (yes/no), and colonic transit time. Stool samples at baseline, end of intervention and after follow-up were obtained in order to be analysed to know about the microbiota. Dietary intake was also recorded at baseline, end of intervention and after follow-up.

Principal subject inclusion criteria: Subjects were recruited if fulfil the Rome III constipation criteria (Mainly hard stools plus stool retention, or pain, or low frequency). Principal subject exclusion criteria: Age under 2 or over 5 years, diapers use, use of laxative during the study and 2 weeks before, use of pre- probiotics or antibiotics during the study and 4 weeks before, organic causes of defecation disorders, other metabolic or renal abnormalities or mental retardation, no parent's command of any local language.

DETAILED DESCRIPTION:
Double-blind, randomised, placebo-controlled parallel group trial (Pilot) Constipated children received two doses of 2g Orafti® inulin-type fructans (OF:IN) or placebo (maltodextrin) for 6 weeks.

Primary outcome was stool consistency. Secondary outcomes were stool frequency and gastrointestinal symptoms. Sample size recruited: twenty-two children, from whom 17 completed the study protocol (nine for the OF:IN and eight for the control group).

ELIGIBILITY:
Inclusion Criteria:

* Two to 5 year-old constipated children with sufficient toilet training.
* To acomplish the Romee I criteria for infants up to 4 yeras. Briefly: have to fulfil at least 2 of the following criteria for at least 1 month:

  1. Two or fewer defecations per week
  2. At least 1 episode per week of incontinence after the acquisition of toileting skills
  3. History of excessive stool retention
  4. History of painful or hard bowel movements
  5. Presence of a large faecal mass in the rectum
  6. History of large-diameter stools that may obstruct the toilet Accompanying symptoms may include irritability, decreased appetite and/or early satiety. Accompanying symptoms disappear immediately following passage of a large stool.

Exclusion Criteria:

* No child's control of defecation (use of diapers).
* No mother's command of any local language.
* Organic causes of defecation disorders incl. Hirschsprung's disease, Spina bifida, hypothyroidism, celiac disease etc.
* Other metabolic or renal abnormalities or mental retardation (Child's mental delay).
* Use of drugs (e.g. antibiotics) and labelled pre- and probiotics influencing gastrointestinal function (4 weeks before run-in, 6 weeks before intervention).
* Use of laxatives in the previous 2 weeks before the beginning of run-in (4 weeks before intervention).

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Escribano, Prof PhD, Principal Investigator — Universitat Rovira i Virgili, IISPV
Locations (1):
- Iispv- Hospital Sant Joan de Reus, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Closa-Monasterolo R, Ferre N, Castillejo-DeVillasante G, Luque V, Gispert-Llaurado M, Zaragoza-Jordana M, Theis S, Escribano J. The use of inulin-type fructans improves stool consistency in constipated children. A randomised clinical trial: pilot study. Int J Food Sci Nutr. 2017 Aug;68(5):587-594. doi: 10.1080/09637486.2016.1263605. Epub 2016 Dec 8. PMID 27931142

RESULTS

PARTICIPANT FLOW:
Groups:
- Inulin-Type Fructans: Orafti inulin-type fructans 2g, twice per day, 6 weeks
  OraftiR inulin-type fructans
Period: Overall Study
Arm/Group | Placebo | Inulin-Type Fructans
Started | 11 | 11
Completed | 9 | 8
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Inulin-Type Fructans | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.03 (0.79) | 3.72 (1.07) | 3.75 (0.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  Spain | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Stool Consistency
Description: Stool consistency was measured according to the Modified Bristol Stool Form Scale for children (from 1 to 5, having lower scores a more hard stool characteristics). Assessed by a continuous daily bowel diary over the following period and in accordance with the Modified Bristol Stool Form Scale for Children. The average consistency from all depositions reported in each follow-up period was obtained for each participant.
Time Frame: 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo: Maltodextrin 2g, twice per day, 6 weeks
Arm/Group | Placebo | Inulin-Type Fructans
Number analyzed (Participants) | 9 | 8
units on a scale | 2.57 (0.58) | 1.63 (0.64)

2. Secondary Outcome: Stool Frequency
Description: Assessed by a continuous daily bowel diary and expressed as average of stools per week
Time Frame: 6 weeks of treatment
Reporting Status: Not Posted

3. Secondary Outcome: Abdominal Pain
Description: Assessed by daily bowel diary and Wong-Baker Faces Pain Rating Scale (scale from 0 to 10 being 0 "no pain" and 10 the "maximum level of pain")
Time Frame: 6 weeks of treatment
Reporting Status: Not Posted

4. Secondary Outcome: Pain During Defecation
Description: as for outcome 3
Time Frame: 6 weeks of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Inulin-Type Fructans
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No